CLINICAL TRIAL: NCT03713489
Title: Platelet Transfusion in HBV-related acute-on Chronic Liver Failure: a Randomized Controlled Study
Brief Title: Platelet Transfusion in HBV-related acute-on Chronic Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Jinjun Chen, Associate Director, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: acute-on-chronic liver failure; platelet; Hepatitis B
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis B | interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet transfusion group (Experimental): Besides standard medical treatment, up to 9 units of platelets will be transfused per protocol within 4 weeks
  Interventions: Procedure: platelet
- standard medical treatment group (No Intervention): standard medical treatment

INTERVENTIONS:
Procedure: platelet — Participants in platelet transfusion group will receive one unit of apheresis platelets transfusion 3 times for the first week after enrollment, then 2 times a week in the following three weeks.
  Arms: Platelet transfusion group

SUMMARY:
Acute-on-chronic liver failure (ACLF) is a syndrome that has recently been recognized as encompassing acute deterioration of liver function in patients with pre-existing chronic liver disease. It is associated with multi-organ failure and a high risk of short-term mortality. Thrombocytopenia is common in ACLF. In addition, the function of platelet is also compromised according to our previous data. The aim of this study is to explore whether platelet transfusion could reduce the short-term mortality rate of HBV-related ACLF. This is a single center, open labeled randomized controlled study. There are two arms. Subjects who is assigned to platelet transfusion group will receive both platelet transfusion (9 times/4 weeks, 1 unit each time) and standard medical treatment. While those in standard medical treatment group will receive standard medical treatment only. The major endpoint is 28-day transplant-free mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old
* Diagnosed with acute-on-chronic liver failure (grade-2) according to EASL-CLIF criteria and grading system.
* Chronic hepatitis B infection.
* ADP inhibition rate ≥70%.

Exclusion Criteria:

* Combined with chronic liver disease other than chronic HBV infection.
* Previous decompensation.
* Intracranial hemorrhage proved by radiological methods, symptoms and physical signs.
* Under anti-platelet or anticoagulants therapy within 4 weeks.
* Esophageal variceal bleeding within 1 week.
* Platelets transfusion within 1 week.
* Hepatocellular carcinoma or other types of malignancies.
* Pregnancy or breastfeeding.
* Severe chronic extra-hepatic disease.
* Comined with situations that researchers considered not suitable for inclusion
* Refusal to sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
28-day transplant-free mortality | 28 days
  whether participant died or not without liver transplantation

SECONDARY OUTCOMES:
transplant-free survival time | 90 days
  survival time without transplation

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatology Unit, Department of Infectious Diseases, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No